CLINICAL TRIAL: NCT03507387
Title: Preventive Intramuscular Phenylephrine in Elective Cesarean Section Under Spinal Anesthesia: A Randomized Controlled Tiral
Brief Title: Preventive Intramuscular Phenylephrine in Elective Cesarean Section Under Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Chao Xu, Principal Investigator, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XYFY2018-KL010-01
Record Dates: First submitted 2018-04-07; First posted 2018-04-25 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Elective Cesarean Section; Spinal Anesthesia
Keywords: Intramuscular; Phenylephrine
MeSH Terms: interventions — Phenylephrine; Saline Solution; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intramuscular phenylephrine group (Experimental): Patients in intramuscular phenylephrine group will receive spinal anesthesia with bupivacaine. 5 mg (1ml) phenylephrine intramuscular injection will be given into the gluteus maximus muscle before anesthesia.1ml of 0.9% normal saline intravenous injection will be given after the subarachnoid injection is completed.
  Interventions: Drug: Phenylephrine; Drug: Normal saline; Drug: Bupivacaine
- Intravenous phenylephrine group (Active Comparator): Patients in intravenous phenylephrine group will receive spinal anesthesia with bupivacaine. 1ml of 0.9% normal saline intramuscular injection will be given into the gluteus maximus muscle before anesthesia.100ug (1ml) phenylephrine intravenous injection will be given after the subarachnoid injection is completed.
  Interventions: Drug: Phenylephrine; Drug: Normal saline; Drug: Bupivacaine
- Placebo group (Placebo Comparator): Patients in intravenous phenylephrine group will receive spinal anesthesia with bupivacaine. 1ml of 0.9% normal saline intramuscular injection will be given into the gluteus maximus muscle before anesthesia. 1ml of 0.9% normal saline intravenous injection will be given after the subarachnoid injection is completed.
  Interventions: Drug: Phenylephrine; Drug: Normal saline; Drug: Bupivacaine

INTERVENTIONS:
Drug: Phenylephrine — 5 mg (1ml) phenylephrine intramuscular injection will be given into the gluteus maximus muscle before anesthesia.100ug (1ml) phenylephrine intravenous injection will be given after the subarachnoid injection is completed .
  Other Names: Metasympatol
Drug: Normal saline — 1ml 0.9% normal saline intramuscular injection will be given into the gluteus maximus muscle before anesthesia and after the subarachnoid injection is completed.
  Other Names: Physiological saline
Drug: Bupivacaine — All patients will receive spinal anesthesia with bupivacaine.
  Other Names: Marcaine

SUMMARY:
Spinal anesthesia is the preferred anesthesia method in cesarean section to provide satisfactory analgesia and muscle relaxant with less impact on respiratory system. However, hypotension often occurred due to the block of sympathetic nerve, causing maternal decline of frontal lobe oxygenation, nausea vomit and the decrease of uteroplacental perfusion. Several measures are used to prevent or treat hypotension caused by spinal anesthesia: prehydration, limb compression, left lateral tilt of operation tables or usage of vasopressors. In the past decade, the most recommended vasopressor to prevent or treat hypotension in spinal anesthesia in cesarean section was phenylephrine, an α-adrenergic receptor, maintaining maternal blood pressure and fetal acid-base state. In clinical work, there are two ways to use phenylephrine : intravenous method with less onset time (several seconds and duration (several minutes) and intramuscular method with longer onset time (10-15 minutes) and duration (1 hour). Many trials demonstrated the protective effect of preventive intravenous phenylephrine on maternal hemodynamics and neonatal acid-base status. However, few trials reported the effect of preventive intramuscular phenylephrine on cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
Hypotension often occurred in parturients undergoing cesarean section in spinal anesthesia. This study aims to determine whether preventive intramuscular phenylephrine can better the fetal acid-base state and maternal hemodynamics.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years to 40 years.
2. Elective cesarean section
3. American Society of Anesthesiologists (ASA) grade from I to Ⅱ, height from 150 cm to 180 cm, BMI<40kg/m2
4. Singleton pregnancy
5. Without pregnancy complications

Exclusion Criteria:

1. Multiple pregnancy
2. Preoperative bradycardia
3. Coagulation dysfunction
4. Parturients with hypertension, diabetes, eclampsia and other pregnancy complications.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Umbilical artery potential of hydrogen (pH) | after the baby is delivered
  detected by a blood gase analyzer

SECONDARY OUTCOMES:
Umbilical venous potential of hydrogen (pH) | after the baby is delivered
  detected by a blood gase analyzer
Umbilical artery base excess | after the baby is delivered
  detected by a blood gase analyzer
Umbilical venous base excess | after the baby is delivered
  detected by a blood gase analyzer
Umbilical artery partial pressure of oxygen (PaO2) | after the baby is delivered
  detected by a blood gase analyzer
Umbilical venous partial pressure of oxygen (PaO2) | after the baby is delivered
  detected by a blood gase analyzer
Umbilical artery partial pressure of carbon dioxide (PaCO2) | after the baby is delivered
  detected by a blood gase analyzer
Umbilical venous partial pressure of carbon dioxide (PaCO2) | after the baby is delivered
  detected by a blood gase analyzer
Umbilical artery lactate | after the baby is delivered
  detected by a blood gase analyzer
Umbilical venous lactate | after the baby is delivered
  detected by a blood gase analyzer
Umbilical artery glucose | after the baby is delivered
  detected by a blood gase analyzer
Umbilical venous glucose | after the baby is delivered
  detected by a blood gase analyzer
Incidence of fetal acidosis | after the baby is delivered
  Umbilical artery pH value<7.20
Incidence of hypotension | intraoperative
  decrease of systolic blood pressure>20% baseline values
Incidence of hypertension | intraoperative
  increase of systolic blood pressure>20% baseline values
Incidence of bradycardia | intraoperative
  heart rate <50 bpm
Incidence of nausea or vomit | intraoperative
  observed by the anesthesiologist

CONTACTS AND LOCATIONS:
Overall Officials: Chao Xu, M.D., Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Foss VT, Christensen R, Rokamp KZ, Nissen P, Secher NH, Nielsen HB. Effect of phenylephrine vs. ephedrine on frontal lobe oxygenation during caesarean section with spinal anesthesia: an open label randomized controlled trial. Front Physiol. 2014 Mar 3;5:81. doi: 10.3389/fphys.2014.00081. eCollection 2014. PMID 24624090
- [Result] Macarthur A, Riley ET. Obstetric anesthesia controversies: vasopressor choice for postspinal hypotension during cesarean delivery. Int Anesthesiol Clin. 2007 Winter;45(1):115-32. doi: 10.1097/AIA.0b013e31802b8d53. No abstract available. PMID 17215703
- [Result] Mon W, Stewart A, Fernando R, Ashpole K, El-Wahab N, MacDonald S, Tamilselvan P, Columb M, Liu YM. Cardiac output changes with phenylephrine and ephedrine infusions during spinal anesthesia for cesarean section: A randomized, double-blind trial. J Clin Anesth. 2017 Feb;37:43-48. doi: 10.1016/j.jclinane.2016.11.001. Epub 2016 Dec 26. PMID 28235526
- [Result] Thomas DG, Robson SC, Redfern N, Hughes D, Boys RJ. Randomized trial of bolus phenylephrine or ephedrine for maintenance of arterial pressure during spinal anaesthesia for Caesarean section. Br J Anaesth. 1996 Jan;76(1):61-5. doi: 10.1093/bja/76.1.61. PMID 8672382
- [Result] Lin FQ, Qiu MT, Ding XX, Fu SK, Li Q. Ephedrine versus phenylephrine for the management of hypotension during spinal anesthesia for cesarean section: an updated meta-analysis. CNS Neurosci Ther. 2012 Jul;18(7):591-7. doi: 10.1111/j.1755-5949.2012.00345.x. PMID 22759268
- [Result] Mohta M, Aggarwal M, Sethi AK, Harisinghani P, Guleria K. Randomized double-blind comparison of ephedrine and phenylephrine for management of post-spinal hypotension in potential fetal compromise. Int J Obstet Anesth. 2016 Aug;27:32-40. doi: 10.1016/j.ijoa.2016.02.004. Epub 2016 Feb 21. PMID 27020488
- [Result] Saravanan S, Kocarev M, Wilson RC, Watkins E, Columb MO, Lyons G. Equivalent dose of ephedrine and phenylephrine in the prevention of post-spinal hypotension in Caesarean section. Br J Anaesth. 2006 Jan;96(1):95-9. doi: 10.1093/bja/aei265. Epub 2005 Nov 25. PMID 16311286
- [Result] Magalhaes E, Goveia CS, de Araujo Ladeira LC, Nascimento BG, Kluthcouski SM. Ephedrine versus phenylephrine: prevention of hypotension during spinal block for cesarean section and effects on the fetus. Rev Bras Anestesiol. 2009 Jan-Feb;59(1):11-20. doi: 10.1590/s0034-70942009000100003. English, Portuguese. PMID 19374211